CLINICAL TRIAL: NCT01418144
Title: Effect of Transversus Abdominis Plane (TAP) Block as Postoperative Pain Management After Laparoscopic Colon Surgery
Brief Title: Effect of Transversus Abdominis Plane (TAP) Block After Laparoscopic Colon Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-HT-2010
Record Dates: First submitted 2011-06-09; First posted 2011-08-16 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Laparoscopic Colon Surgery
MeSH Terms: interventions — Dental Occlusion; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transversus abdominis plane (TAP) block (Experimental): Transversus abdominis plane (TAP) block with ropivacaine
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- Block with saline (Placebo Comparator): Bilateral placement of 20 ml of saline 0,9% in the transversus abdominis plane
  Interventions: Procedure: Placebo TAP block

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — Bilateral UL-guided TAP block with 20 ml of ropivacaine 0,5%
  Other Names: Naropin
  Arms: Transversus abdominis plane (TAP) block
Procedure: Placebo TAP block — Bilateral placement of 20 ml of saline 0,9% in the transversus abdominis plane
  Other Names: Placebo block
  Arms: Block with saline

SUMMARY:
The purpose of this study is to investigate the effectiveness of Transversus Abdominis Plane (TAP) block as a part of a multimodal postoperative pain management after laparoscopic surgery on colon.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80
* BMI 18 - 40
* ASA 1 - 3
* Written consent
* Can cooperate

Exclusion Criteria:

* Mb Chron and Collitis Ulcerosa
* Drug and alcohol abuse
* Pregnancy
* Consumption of opioids
* Drug allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain during cough | 6 hours
  VAS-pain score

SECONDARY OUTCOMES:
Pain during rest | 1,2,4,6,12 and 24 hours
  VAS-pain score at rest
Total opioid consumption | 0-24 hours
  Opioid consumption via PCA-pump.
Postoperative nausea and vomiting | 1,2,4,6,12,18 and 24 hours
  Nausea score 0-3 No. of vomits

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev University Hospital, Department of anaesthesia, Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Torup H, Hansen EG, Bogeskov M, Rosenberg J, Mitchell AU, Petersen PL, Mathiesen O, Dahl JB, Moller AM. Transversus abdominis plane block after laparoscopic colonic resection in cancer patients: A randomised clinical trial. Eur J Anaesthesiol. 2016 Oct;33(10):725-30. doi: 10.1097/EJA.0000000000000510. PMID 27487909